CLINICAL TRIAL: NCT00645736
Title: Study of Acquired Viral Mutations in Chronic Hepatitis B Patients on Antihepadnaviral Therapy
Brief Title: CHARM: Chronic Hepatitis B Antihepadnaviral Resistance Mutation Study
Acronym: CHARM
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-AU-103-0185
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Single cohort
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study has the aim of describing viral mutation profiles in patients diagnosed with chronic hepatitis B receiving antihepadnaviral therapy.

DETAILED DESCRIPTION:
This is a naturalistic cross-sectional study of chronic hepatitis B subjects receiving nucleoside or nucleotide antihepadnaviral therapy.

It is anticipated approximately 800 subjects will be recruited at 20 Australian sites. Data will be collected on the study subjects and analyses performed to describe factors contributing to the emergence of viral mutations in Australian patients with chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over
* Provided informed consent
* Diagnosis of chronic hepatitis B (HBsAg documented for at least 6 months)
* Currently prescribed antihepadnaviral therapy (including, but not limited to: lamivudine, adefovir, entecavir, tenofovir or telbivudine) for chronic hepatitis B management
* Been taking current antihepadnaviral therapy for at least 6 months prior to recruitment
* Negative tests for HIV Ab, Hepatitis C Ab and Hepatitis D Ab within the previous 2 years

Exclusion Criteria:

* Known or suspected co-infection with HIV, Hepatitis C or Hepatitis D
* Concomitant immunosuppression / immunomodulatory therapies
* Diagnosis of hepatocellular carcinoma where anticipated life expectancy is less than 6 months
* Current participation in an interventional, blinded, pharmaceutical industry-sponsored clinical trial
* Current Child Pugh class C classification (current Child Pugh score > 9)
* Other known or suspected cause of chronic liver disease
* Any other reason that, in the investigator's opinion, participation in the study would not be in the participant's best interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diagnosis of chronic hepatitis B who have been prescribed antihepadnaviral therapy for at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 788 (Actual)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Descriptive statistics for clinical and viral characteristics of the study population | Single timepoint (blood draw)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Wraight, Study Director — Gilead Sciences Pty Ltd
Locations (1):
- Gilead Sciences Pty Ltd, East Melbourne, Victoria, Australia